CLINICAL TRIAL: NCT03456141
Title: Prospective, Observational Study With a Multimodal Analgesic Protocol to Moderate Acute Pain After Third Molar Surgery
Brief Title: Multimodal Analgesic Protocol to Moderate Acute Pain
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0047
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-12

CONDITIONS: Pain, Post-operative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: third molar surgery — The patient is asked to complete the diary each post-surgery day for 14 days. Recovery is organized into three QOL domains: lifestyle, oral function, and pain.

SUMMARY:
With a prospective, observational study assess post-surgery pain levels and patient's use of opioids and other analgesic drugs to moderate pain following third molar surgery.

DETAILED DESCRIPTION:
SPECIFIC AIMS Using the UNC surgery clinic multi-modal protocol of drugs/dosages to control acute pain after third molar surgery assess each post-surgery day(PSD) the patient reported

1. pain levels post-surgery as recorded by Likert-type and Gracely scales
2. quality of life(QOL) outcomes for lifestyle and oral function
3. number of opioid doses taken by subject-patients
4. number of NSAID and acetaminophen doses taken by subject-patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II At least two lower 3rd molars scheduled for removal

Exclusion Criteria:

* Patient being treated for opioid addiction/abuse including having Rx for suboxone, methadone

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients scheduled for surgery at UNC oral and maxillofacial surgery clinic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The impact of the surgery on the patient's post-surgery pain. | 14 days
  Likert scales for average pain and worst pain are assessed with 7-point scales with verbal anchors of "no pain" and "worst pain imagined".
  Recovery for pain on the Likert scales is defined as the number of PSD until the patient reports a score of 1 or 2 on the 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Reside, DMD, Principal Investigator — UNC oral and maxillofacial surgery
Locations (1):
- University of North Carolina School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No